CLINICAL TRIAL: NCT05914753
Title: A Prospective Clinical Study Evaluating Xihuang Pill to Improve the Efficacy of Neoadjuvant Chemotherapy for Breast Cancer
Brief Title: Evaluating Xihuang Pill to Improve the Efficacy of Neoadjuvant Chemotherapy for Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Xuli Meng, Chief physician, Zhejiang Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHWBC
Record Dates: First submitted 2023-06-04; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Chemotherapy Effect
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Experimental group: Epirubicin :90 mg/m2, D1, q3W; Cyclophosphamide :600 mg/m2, D1, q3W; Xihuang Pill：3g po bid，4 cycles, Follow Docetaxel :100 mg/m2, D1, q3W；Xihuang Pill：3g po bid，4 cycles
  Interventions: Drug: Epirubicin, Cyclophosphamide, Xihuang Pill, Docetaxel
- Control group (Placebo Comparator): Control group: Epirubicin :90 mg/m2, D1, q3W; Cyclophosphamide :600 mg/m2, D1, q3W，4 cycles, Follow Docetaxel :100 mg/m2, D1, q3W，4 cycles
  Interventions: Drug: Epirubicin, Cyclophosphamide, Docetaxel

INTERVENTIONS:
Drug: Epirubicin, Cyclophosphamide, Xihuang Pill, Docetaxel — Epirubicin :90 mg/m2, D1, q3W; Cyclophosphamide :600 mg/m2, D1, q3W; Xihuang Pill：3g po bid，4 cycles, Follow Docetaxel :100 mg/m2, D1, q3W；Xihuang Pill：3g po bid，4 cycles
  Arms: Experimental group
Drug: Epirubicin, Cyclophosphamide, Docetaxel — Epirubicin :90 mg/m2, D1, q3W; Cyclophosphamide :600 mg/m2, D1, q3W，4 cycles, Follow Docetaxel :100 mg/m2, D1, q3W，4 cycles
  Arms: Control group

SUMMARY:
Evaluate the effectiveness of Xihuang Pill in improving the efficacy of neoadjuvant chemotherapy for breast cancer

DETAILED DESCRIPTION:
1. To evaluate the safety and effectiveness of Xihuang Pill in improving the efficacy of neoadjuvant chemotherapy for breast cancer under the condition of widespread use.
2. To provide data support for improving the efficacy of neoadjuvant chemotherapy for clinical breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy of breast mass was performed under ultrasound-guided treatment before neoadjuvant chemotherapy, and the diagnosis of breast cancer was confirmed pathologically, followed by immunohistochemical examination. Pathological sections before and after neoadjuvant chemotherapy were jointly diagnosed by 3 or more senior pathologists, and there were consistent definite conclusions.
2. Have detailed and complete clinicopathological data;
3. Diagnosis data of TCM syndrome type;
4. No biopsy-confirmed lymph node metastasis;
5. No serious systemic disease, able to tolerate neoadjuvant chemotherapy and surgical treatment;
6. At least 4 cycles of neoadjuvant chemotherapy were completed, and the efficacy of chemotherapy was evaluated at the end of chemotherapy and after surgery;
7. Under the guidance of doctors, take Xihuang pills in a standardized way throughout the whole process and review regularly;
8. The patient did not receive any antitumor therapy drugs associated with the tumor prior to neoadjuvant chemotherapy;
9. All patients were newly diagnosed

Exclusion Criteria:

1. Concurrent malignant tumors of other sites;
2. Patients with distant metastasis
3. Male breast cancer
4. Patients who did not receive full-course standardized neoadjuvant chemotherapy;
5. Lost contact or dropped out of the study, unable to follow up;
6. Inability to tolerate chemotherapy responses;
7. Intolerant to Xihuang Wan and unable to take it;
8. The patient has strong side effects of chemotherapy and cannot tolerate chemotherapy drugs;
9. Inflammatory breast cancer, bilateral breast cancer, paget's disease and other special types of breast cancer;
10. Various other possible influences.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | six months
  Pathological complete response

CONTACTS AND LOCATIONS:
Overall Officials: Xuli Meng, Study Chair — Zhejiang Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No
After preliminary results are available, it is advisable to decide whether to share them with other researchers.